CLINICAL TRIAL: NCT00820222
Title: A Randomized, Multicentre, Open-Label, Phase III Study of Lapatinib Plus Capecitabine Versus Trastuzumab Plus Capecitabine in Patients With Anthracycline- or Taxane-Exposed ErbB2-Positive Metastatic Breast Cancer
Brief Title: Lapatinib Plus Capecitabine Versus Trastuzumab Plus Capecitabine in ErbB2 (HER2) Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111438
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Metastases, Brain
Keywords: ErbB2; HERCEPTIN; XELODA; ErbB1; TYKERB; metastatic breast cancer; trastuzumab; breast cancer; capecitabine; lapatinib; brain metastases; HER2 positive; TYVERB
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms | interventions — Capecitabine; Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lapatinib plus capecitabine (Experimental): Lapatinib 1250 mg once daily and capecitabine 2000mg/m2/day, days 1-14, every 21 days
  Interventions: Drug: capecitabine; Drug: lapatinib
- Trastuzumab plus capecitabine (Active Comparator): trastuzumab loading dose of 8mg/kg followed by 6mg/kg q3weekly infusions, and capecitabine 2500mg/m2/day, days 1-14, every 21 days
  Interventions: Drug: capecitabine; Drug: trastuzumab

INTERVENTIONS:
Drug: capecitabine — oral medication; daily dose divided into morning and evening dose and taken for 14 days of 21 day cycle
Drug: lapatinib — oral medication; daily dose taken once a day
  Arms: Lapatinib plus capecitabine
Drug: trastuzumab — infusion therapy; loading dose of 8mg/kg, followed by 6mg/kg given every 3 weeks
  Arms: Trastuzumab plus capecitabine

SUMMARY:
This open label study was designed to evaluate Lapatinib effect on incidence of brain metastases in ErbB2 (HER2) positive metastatic breast cancer patients exposed to prior taxanes or anthracyclines.

DETAILED DESCRIPTION:
The study was terminated based on the IDMC recommendation in 2012, collection of efficacy outcome measures was discontinued and all primary and secondary outcome measures were reported in 2012.

An amendment protocol allowed subjects who were on study treatment to enroll in a Long Term Follow Up (LTFU) phase if they had evidence of clinical benefit but no local access to standard of care treatments. Subjects received study treatment until disease progression, unacceptable toxicity, or subject withdrawal. In LTFU only Adverse Events data were collected. For the LTFU the Outcome Measure "Number of participants with the indicated Grade 3 or Grade 4 Adverse Events (AEs) occurring in >=2% of participants in either treatment arm" and "Adverse Events" were updated.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 18 years old;
* ECOG Performance Status 0-2;
* Histologically or cytologically confirmed HER2-positive invasive breast cancer, with Stage IV disease;
* Prior treatment with taxanes or anthracyclines is required;
* Prior treatment with other chemotherapeutic agents, trastuzumab, endocrine and radiation therapy is permitted;
* Baseline LVEF ≥ 50% and not lower than the institutional lower limit of normal;
* Concurrent treatment with bisphosphonates is permitted, however treatment must be initiated prior to the first dose of study therapy;
* Able to swallow and retain oral medications;
* Women with potential to have children must be willing to practice acceptable methods of birth control during the study;
* Normal organ and marrow function.

Exclusion Criteria:

* History and/or current evidence of CNS metastases. Baseline MRI scan by Independent Reviewer to confirm no brain mets;
* Concurrent treatment with an investigational agent or participation in another treatment clinical trial;
* Prior therapy with lapatinib or an ErbB2 inhibitor other than trastuzumab (including but not limited to trastuzumab-DM1 and neratinib) and capecitabine;
* Known DPD deficiency;
* Concurrent chemotherapy, radiation therapy, immunotherapy, biologic therapy, or hormonal therapy for treatment of cancer;
* History of allergic reactions attributed to compounds chemically related to lapatinib (quinazolines), capecitabine, fluorouracil or any excipients;
* Concomitant use of CYP3A4 inhibitors or inducers;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel;
* History of immediate or delayed hypersensitivity reaction to gadolinium contrast agents, or other contraindication to gadolinium contrast and other known contraindication to MRI;
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the patient's safety or compliance to study procedures;
* have acute or currently active/requiring anti-viral therapy hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease);
* Any on-going toxicity from prior anti cancer therapy except alopecia;
* Active cardiac disease;
* Uncontrolled infection;
* History of other malignancy, unless curatively treated with no evidence of disease for at least 5 years, subjects with adequately treated DCIS or LCIS, adequately treated non-melanoma skin cancer or curatively treated in-situ cancer of the cervix are eligible;
* Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of protocol treatment;
* Pregnant or lactating females.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2009-04-14 (Actual); Primary Completion 2012-06-11 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (145):
- United States (17):
  - Novartis Investigative Site, Goodyear, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Greenbrae, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Santa Barbara, California
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Coral Springs, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Warrenville, Illinois
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Voorhees Township, New Jersey
  - Novartis Investigative Site, Durham, North Carolina
- Belgium (3):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Sint-Niklaas
- Novartis Investigative Site, Aarhus, Denmark
- France (14):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Dechy
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Saint-Grégoire
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Vannes
- Germany (27):
  - Novartis Investigative Site, Ravensburg, Baden-Wurttemberg
  - Novartis Investigative Site, Eggenfelden, Bavaria
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Landshut, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Nuremberg, Bavaria
  - Novartis Investigative Site, Rosenheim, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Potsdam, Brandenburg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Wiesbaden, Hesse
  - Novartis Investigative Site, Bottrop, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Duisburg, North Rhine-Westphalia
  - Novartis Investigative Site, Goch, North Rhine-Westphalia
  - Novartis Investigative Site, Herne, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Witten, North Rhine-Westphalia
  - Novartis Investigative Site, Würselen, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Speyer, Rhineland-Palatinate
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Brandenburg
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Hamburg
- Greece (6):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, N. Kifisia, Athens
  - Novartis Investigative Site, Neo Faliro
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Peiraius
  - Novartis Investigative Site, Thessaloniki
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Tatabánya
  - Novartis Investigative Site, Veszprém
- Italy (14):
  - Novartis Investigative Site, Bologna, Emilia-Romagna
  - Novartis Investigative Site, Meldola (FC), Emilia-Romagna
  - Novartis Investigative Site, Rimini, Emilia-Romagna
  - Novartis Investigative Site, Udine, Friuli Venezia Giulia
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Monza, Lombardy
  - Novartis Investigative Site, Treviglio (BG), Lombardy
  - Novartis Investigative Site, Novara, Piedmont
  - Novartis Investigative Site, Fermo (AP), The Marches
  - Novartis Investigative Site, Trento, Trentino-Alto Adige
  - Novartis Investigative Site, Lido Di Camaiore (LU), Tuscany
  - Novartis Investigative Site, Pisa, Tuscany
  - Novartis Investigative Site, Perugia, Umbria
  - Novartis Investigative Site, Varese
- Poland (8):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bytom
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Wroclaw
- Russia (15):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Moscow Region
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Obninsk
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Veliky Novgorod
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Vsevolozhsk
- Spain (13):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Cáceres
  - Novartis Investigative Site, Hospitalet de Llobregat (Barcelona)
  - Novartis Investigative Site, Jerez (Cadiz)
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Torrevieja (Alicante)
  - Novartis Investigative Site, Valencia
- Sweden (4):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Vaxjo
  - Novartis Investigative Site, Västerås
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Songkhla
- United Kingdom (16):
  - Novartis Investigative Site, Edinburgh, Midlothian
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Aberdeen
  - Novartis Investigative Site, Burton-on-Trent
  - Novartis Investigative Site, Cottingham, Hull
  - Novartis Investigative Site, Huddersfield
  - Novartis Investigative Site, Ipswich
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Maidstone
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Peterborough
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Shrewsbury
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Wolverhampton
  - Novartis Investigative Site, Worthing

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pivot X, Manikhas A, Zurawski B, Chmielowska E, Karaszewska B, Allerton R, Chan S, Fabi A, Bidoli P, Gori S, Ciruelos E, Dank M, Hornyak L, Margolin S, Nusch A, Parikh R, Nagi F, DeSilvio M, Santillana S, Swaby RF, Semiglazov V. CEREBEL (EGF111438): A Phase III, Randomized, Open-Label Study of Lapatinib Plus Capecitabine Versus Trastuzumab Plus Capecitabine in Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer. J Clin Oncol. 2015 May 10;33(14):1564-73. doi: 10.1200/JCO.2014.57.1794. Epub 2015 Jan 20. PMID 25605838

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib Plus Capecitabine: Participants received a daily dose of 5 tablets of lapatinib (1250 milligrams [mg]) at approximately the same time every day, either 1 hour (or more) before breakfast or 1 hour (or more) after breakfast. Participants also received capecitabine 2000 mg per meters squared (mg/m^2) per day (divided and administered orally twice daily, 12 hours apart), for 14 days, every 21 days. Capecitabine was taken with food or within 30 minutes after food. Participants received study medication until disease progression, unacceptable toxicity, or participant withdrawal.
- Trastuzumab Plus Capecitabine: Participants received an intravenous (IV) infusion of trastuzumab 8 mg/kilogram (kg) on Day 1, followed by a 6 mg/kg infusion every 3 weeks. Participants also received capecitabine 2500 mg/m^2 per day (divided and administered orally twice daily, 12 hours apart), for 14 days, every 21 days. Capecitabine was taken with food or within 30 minutes after food. Participants received study medication until disease progression, unacceptable toxicity, or participant withdrawal.
Period: Overall Study
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Started | 271 | 269
Completed | 95 | 79
Not Completed | 176 | 190
Not completed — Lost to Follow-up | 10 | 9
Not completed — Withdrawal by Subject | 19 | 21
Not completed — Physician Decision | 93 | 88
Not completed — Sponsor Terminated Study | 43 | 65
Not completed — Unkown | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Trastuzumab Plus Capecitabine: Participants received an IV infusion of trastuzumab 8 mg/kg on Day 1, followed by a 6 mg/kg infusion every 3 weeks. Participants also received capecitabine 2500 mg/m^2 per day (divided and administered orally twice daily, 12 hours apart), for 14 days, every 21 days. Capecitabine was taken with food or within 30 minutes after food. Participants received study medication until disease progression, unacceptable toxicity, or participant withdrawal.
- Total: Total of all reporting groups
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine | Total
Number analyzed (Participants) | 271 | 269 | 540
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (10.23) | 55.8 (10.26) | 54.6 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 271 | 269 | 540
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European | 266 | 260 | 526
  White - Arabic/North African Heritage | 0 | 1 | 1
  African American/African Heritage | 1 | 1 | 2
  Asian - Central/South Asian Heritage | 1 | 1 | 2
  Asian - East Asian Heritage | 1 | 2 | 3
  Asian - South East Asian Heritage | 2 | 3 | 5
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Central Nervous System (CNS) Metastases (as Assessed by Independent Review) as the Site of First Relapse
Description: CNS relapse is defined as the appearance of >=1 enhancing lesion measuring >=6 millimeters (mm) on T1Weighted (T1W) Magnetic Resonance Imaging (MRI) without CNS symptoms that were considered to be unequivocal based on all relevant radiological features (e.g., associated T2W signal abnormality); the appearance of any enhancing lesion on T1W MRI with CNS symptoms; unequivocal finding of leptomeningeal disease (defined as the dissemination of cancer throughout the spinal fluid), with or without symptoms; and unequivocal finding of multifocal intraparenchymal lesions with or without symptoms. In the event of the appearance of a <6 mm lesions(s) without CNS lesions, or equivocal findings potentially suggesting leptomeningeal disease, these findings were followed with a subsequent scan within 6 weeks. If unequivocal progression was determined with the subsequent scan and/or CNS symptoms occurred, then CNS relapse crieria were met.
Time Frame: From randomization until disease progression, death, or discontinuation from the study (average of 10 months). Cut-off 11-Jun-2012
Population: Modified Intent-to-Treat (M-ITT) Population: all participants who were randomized to study treatment regardless of whether or not treatment was administered and who had no Baseline CNS metastases per Independent Review Committee (IRC) assessment
Measure: Number; unit: participants
Groups:
- Lapatinib Plus Capecitabine: Participants received a daily dose of 5 tablets of lapatinib (1250 mg) at approximately the same time every day, either 1 hour (or more) before breakfast or 1 hour (or more) after breakfast. Participants also received capecitabine 2000 mg/m^2) per day (divided and administered orally twice daily, 12 hours apart), for 14 days, every 21 days. Capecitabine was taken with food or within 30 minutes after food. Participants received study medication until disease progression, unacceptable toxicity, or participant withdrawal.
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 251 | 250
participants | 8 | 12
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine vs Trastuzumab Plus Capecitabine; Test type: Superiority or Other; p = 0.360, Odds Ratio; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.26 to 1.63] — The Odds Ratio is based on a logistic regression model. The P-value for the test of Odds Ratio is 1

2. Secondary Outcome: Progression Free Survival (PFS), as Assessed by the Investigator
Description: PFS is defined as the interval between the date of randomization and the earliest date of progressive disease (PD), or death due to any cause. PD is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, compared with the smallest sum LD recorded since the treatment started, or the appearance of 1 or more new lesions based on investigator assessment of both CNS and non-CNS for response.
Time Frame: as for outcome 1
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to study treatment regardless of whether or not treatment was administered
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 271 | 269
months | 6.60 [5.72 to 8.11] | 8.05 [6.14 to 8.90]
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine vs Trastuzumab Plus Capecitabine; Test type: Superiority; p = 0.021, Log Rank; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [1.04 to 1.64] — A HR > 1 indicates a higher risk for lapatinib+capecitabine compared with trastuzumab+capecitabine

3. Secondary Outcome: Time to First CNS Progression, Defined as the Time From Randomization Until the Date of Documented CNS Progression as the First Site of Relapse
Description: CNS relapse is defined as the appearance of >=1 enhancing lesion measuring >=6 mm on T1W MRI without CNS symptoms that were considered to be unequivocal based on all relevant radiological features (e.g., associated T2W signal abnormality); the appearance of any enhancing lesion on T1W MRI with CNS symptoms; unequivocal finding of leptomeningeal disease (defined as the dissemination of cancer throughout the spinal fluid), with or without symptoms; and unequivocal finding of multifocal intraparenchymal lesions with or without symptoms. In the event of the appearance of a <6 mm lesions(s) without CNS lesions, or equivocal findings potentially suggesting leptomeningeal disease, these findings were followed with a subsequent scan within 6 weeks. If unequivocal progression was determined with the subsequent scan and/or CNS symptoms occurred, then CNS relapse crieria were met.
Time Frame: From randomization until the date of documented CNS progression (average of 10 months). Cut-off 11-Jun-2012
Population: M-ITT Population. Only those participants who had no Baseline CNS metastases and who had CNS progression by radiographic confirmation (per Response Evaluation Criteria in Solid Tumors, 1.0: a 20% increase in the sum of the longest diameter [LD] of target lesions or the appearance of >=1 new lesions) were included in this analysis.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 8 | 12
months | 8.2 (6.78) | 6.7 (6.94)

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death due to any cause or to the date of censor. In the absence of confirmation of death, survival time was to be censored at the time of the last investigator contact.
Time Frame: From randomization until death due to any cause (average of 10 months). Cut-off 11-Jun-2012
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 271 | 269
months | 22.7 [19.5 to NA] — The upper limit of the 95% confidence interval could not be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI. | 27.3 [23.7 to NA] — The upper limit of the 95% confidence interval could not be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI.
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine vs Trastuzumab Plus Capecitabine; Test type: Superiority; p = 0.095, Log Rank; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.95 to 1.90] — A HR > 1 indicates a higher risk for lapatinib+capecitabine compared with trastuzumab+capecitabine

5. Secondary Outcome: Number of Participants With Overall Response (OR), as Assessed by the Investigator
Description: OR is defined as the number of participants with either a confirmed complete response (CR; disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of the LD of the target lesions, compared with the baseline sum LD). CR and PR were assessed per Response Evaluation Criteria in Solid Tumors (RECIST). To be assigned a status of PR or CR, a confirmatory disease assessment was to be performed 28 days (4 weeks) or greater after the criteria for response were first met. In addition, a bone scan must have been obtained to rule out the presence of new bone lesions or progression of existing bone lesions, even if the participant had no bone lesions present at Baseline. If a bone scan was performed at the time of initial response or near the time of response, the bone scan did not need to be repeated.
Time Frame: as for outcome 1
Population: ITT Population. Only those participants enrolled under protocol amendment 3 were required to have PR or CR confirmation. Those participants enrolled under protocol amendments 1 and 2 were considered to have a "confirmed" response at the time of the first PR or CR regardless of follow-up scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 271 | 269
Participants
  CR | 8 | 12
  PR | 65 | 73
  Overall Response (CR+PR) | 73 | 85
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine vs Trastuzumab Plus Capecitabine; Comparison for Overall Response (CR+PR); Test type: Superiority; p = 0.2731, Fisher Exact; Odds Ratio (OR) = 0.7984, 95% CI 2-sided [0.5407 to 1.1771]

6. Secondary Outcome: Number of Participants With Clinical Benefit (CB)
Description: CB is defined as the number of participants with evidence of confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of the LD of the target lesions, compared with the baseline sum LD) at any time or stable disease (SD, neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD [defined as at least a 20% increase in the sum of the LD of target lesions, compared with the smallest sum LD recorded since the treatment started, or the appearance of 1 or more new lesions] based on investigator assessment), for at least 24 weeks.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 271 | 269
Participants
  CR | 8 | 12
  PR | 65 | 73
  SD >= 24 weeks | 39 | 33
  Clinical Benefit (CR + PR + SD >= 24 weeks) | 112 | 118
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine vs Trastuzumab Plus Capecitabine; Comparison for Clinical Benefit; Test type: Superiority; p = 0.6106, Fisher Exact; Odds Ratio (OR) = 0.9016, 95% CI 2-sided [0.6315 to 1.2866]

7. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the first documented evidence of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of the LD of the target lesions, compared with the baseline sum LD) until the first documented sign of PD (at least a 20% increase in the sum of the LD of target lesions, compared with the smallest sum LD recorded since the treatment started, or the appearance of 1 or more new lesions) or death due to breast cancer. In the absence of confirmation of death, survival time was to be censored at the time of the last investigator contact.
Time Frame: From the time of the first documented confirmed complete or partial response until disease progression or death, if sooner (average of 10 months). Cut-off 11-Jun-2012
Population: ITT Population. Only those participants with CR or PR showing PD or death due to breast cancer were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 73 | 85
months | 6.2 [5.3 to 10.6] | 8.4 [6.0 to 21.6]

8. Secondary Outcome: Number of Participants With CNS Progression at Any Time
Description: CNS progression was documented by a brain scan and was indicated by the investigator on the follow-up electronic Case Report Form. CNS relapse is defined as the appearance of >=1 enhancing lesion measuring >=6 mm on T1W MRI without CNS symptoms that were considered to be unequivocal based on all relevant radiological features (e.g., associated T2W signal abnormality); the appearance of any enhancing lesion on T1W MRI with CNS symptoms; unequivocal finding of leptomeningeal disease, with or without symptoms; and unequivocal finding of multifocal intraparenchymal lesions with or without symptoms. In the event of the appearance of a <6 mm lesions(s) without CNS lesions, or equivocal findings potentially suggesting leptomeningeal disease, these findings were followed with a subsequent scan within 6 weeks. If unequivocal progression was determined with the subsequent scan and/or CNS symptoms occurred, then CNS relapse crieria were met.
Time Frame: From the time of randomization until death due to any cause (average of 10 months). Cut-off 11-Jun-2012
Population: M-ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 251 | 250
participants | 17 | 15

9. Secondary Outcome: Number of Participants With Qualitative and Quantitative Toxicities
Description: Qualitative and quantitative toxicities were measured as AEs. See the outcome measure entitled "Number of participants with the indicated Grade 3 or Grade 4 Adverse Events (AEs) occurring in >=2 participants in either treatment arm" and the AE module of this results summary for a list of AEs occurring in the study. An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: From the first dose of study medication until 30 days after the last dose of study treatment (average of 10 months)
Population: Safety Population
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants Expressing Glucocorticoid Receptor, Phosphatase and Tensin Homolog (PTEN), Phosphatidylinositide 3-kinase (PI3K)/AKT, Protein 53 (P53), Insulin-like Growth Factor-1 (IGF-1), and Genes Involved in Cell Cycle Regulation
Description: Because the study terminated early, pharmacogenetic and biomarker analyses were not performed.
Time Frame: Baseline
Population: ITT Population
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Adverse Events (AEs) Occurring in >=2% of Participants in Either Treatment Arm
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The Investigator assessed whether the AE was related to study drug. AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0=No AE or within normal limits; 1=Mild AE; 2=Moderate AE; 3=Severe and undesirable AE; 4=Life-threatening or disabling AE; 5=Death related to AE.
Time Frame: From the first dose of study medication until 30 days after the last dose of study treatment (average of 10 months).
Population: Safety Population: all participants in the ITT Population who received at least one dose of investigational product, based on the actual treatment received if this differed from that to which the participant was randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
Number analyzed (Participants) | 270 | 267
Participants
  Palmar-plantar erythrodysaesthesia syndrome | 29 | 45
  Diarrhoea | 19 | 22
  Aspartate aminotransferase increased | 11 | 4
  Neutropenia | 9 | 18
  Asthenia | 9 | 6
  Fatigue | 7 | 4
  Alanine aminotransferase increased | 4 | 6
  Hypokalaemia | 3 | 11

ADVERSE EVENTS:
Time Frame: From randomization until up to and including 30 days after the last dose of study treatment (up to 7 years post randomization)
Arm/Group | Lapatinib Plus Capecitabine | Trastuzumab Plus Capecitabine
All-Cause Mortality (participants affected / at risk) | 12/270 | 3/267
Serious Adverse Events (participants affected / at risk) | 41/270 | 51/267
Other Adverse Events (participants affected / at risk) | 241/270 | 236/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Capecitabine (N=270) | Trastuzumab Plus Capecitabine (N=267)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
Biliary colic (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 2
Thrombosis (Vascular disorders) | 0 | 2
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Capecitabine (N=270) | Trastuzumab Plus Capecitabine (N=267)
Anaemia (Blood and lymphatic system disorders) | 22 | 27
Leukopenia (Blood and lymphatic system disorders) | 11 | 21
Neutropenia (Blood and lymphatic system disorders) | 38 | 44
Abdominal pain upper (Gastrointestinal disorders) | 21 | 16
Diarrhoea (Gastrointestinal disorders) | 125 | 107
Dyspepsia (Gastrointestinal disorders) | 21 | 19
Nausea (Gastrointestinal disorders) | 82 | 50
Stomatitis (Gastrointestinal disorders) | 16 | 23
Vomiting (Gastrointestinal disorders) | 35 | 27
Asthenia (General disorders) | 46 | 45
Fatigue (General disorders) | 26 | 33
Mucosal inflammation (General disorders) | 21 | 27
Pyrexia (General disorders) | 19 | 25
Hyperbilirubinaemia (Hepatobiliary disorders) | 35 | 26
Alanine aminotransferase increased (Investigations) | 34 | 35
Aspartate aminotransferase increased (Investigations) | 33 | 30
Blood alkaline phosphatase increased (Investigations) | 17 | 11
Blood bilirubin increased (Investigations) | 19 | 9
Decreased appetite (Metabolism and nutrition disorders) | 28 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 9
Headache (Nervous system disorders) | 15 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 18
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 21 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 142 | 160
Rash (Skin and subcutaneous tissue disorders) | 66 | 21

LIMITATIONS AND CAVEATS:
In 2012 enrollment was stopped and collection of efficacy outcome measures discontinued. Subjects were allowed to enroll in a Long Term Follow Up to provide continued access in which only AE information was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.